CLINICAL TRIAL: NCT00394121
Title: Long-term Open-label Safety Study With SkyePharma FlutiForm HFA pMDI (100/10 µg and 250/10 µg) in Adult and Adolescent Patients With Asthma
Brief Title: New Combination Inhaler (FlutiForm HFA MDI 100/10 µg and 250/10 µg) in Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKY2028-3-003
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Asthma
Keywords: Asthma; Fluticasone Propionate; Formoterol Fumarate; Pressurized metered does inhaler; Hydrofluoroalkane; Mild to moderate-severe asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Formoterol Fumarate

INTERVENTIONS:
Drug: Fluticasone propionate/formoterol fumarate

SUMMARY:
The purpose of this study is to evaluate the long-term safety of the fixed combination asthma drug FlutiForm HFA MDI (containing fluticasone propionate and formoterol fumarate) in adult and adolescent patients with mild to moderate-severe asthma.

ELIGIBILITY:
Ages eligible for study: 12 years and above; genders eligible for study: both; prior steroid use: steroid-requiring.

Inclusion Criteria:

* History of asthma for at least 12 months.
* Documented use of inhaled corticosteriod for at least 4 weeks prior to Screening Visit Demonstrate FEV-1 of 40-80% of predicted normal values at Screening and Baseline Visit.
* Documented reversibility of 15% within 6 months of Screening Visit or at Screening Visit (15% increase from pre-FEV-1 levels following albuterol inhalation).
* Symptoms of Asthma during Run-in.
* Females of childbearing potential must have a negative urine pregnancy test at Screening and Baseline Visits. Females are eligible only if they are not pregnant or lactating and are either sterile or using acceptable methods of contraception.
* Must otherwise be healthy.
* Provide written informed consent. Wishes of minors must be respected.

Exclusion Criteria:

* Life-threatening asthma within past year or during Run-in Period.
* History of systemic corticosteroid medication within 3 months before Screening Visit.
* History of omalizumab use within the past 6 months.
* History of leukotriene receptor antagonist use, e.g., montelukast, within the past week.
* Current evidence of history of any clinically significant disease or abnormality including uncontrolled hypertension, uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia.
* Upper or lower respiratory infection within 4 weeks prior to Screening Visit or during Run-in Period.
* Significant, non-reversible, pulmonary disease (e.g., chronic obstructive pulmonary disease [COPD], cystic fibrosis, bronchiectasis).
* Known Human Immunodeficiency Virus (HIV)-positive status.
* Smoking history equivalent to "10 pack years".
* Current smoking history within 12 months prior to Screening Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Long-term safety after twice daily treatment with FlutiForm HFA MDI over 12 months.

SECONDARY OUTCOMES:
Long-term efficacy after twice daily treatment with FlutiForm HFA MDI over 12 months.

CONTACTS AND LOCATIONS:
Locations (28):
- Germany (5):
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Mainz
  - Research Site, Rüdersdorf
  - Research Site, Solingen
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Wroclaw
- Research Site, Bucharest, Romania
- United Kingdom (12):
  - Research Site, Birmingham
  - Research Site, Carrickfergus
  - Research Site, Chippenham
  - Research Site, Cottingham
  - Research Site, Coventry
  - Research Site, Downpatrick
  - Research Site, Heywood
  - Research Site, Manchester
  - Research Site, Sheffield
  - Research Site, Solihull
  - Research Site, Sunbury-on-Thames
  - Research Site, Swindon Wilts

REFERENCES:
- [Derived] Mansur AH, Kaiser K. Long-term safety and efficacy of fluticasone/formoterol combination therapy in asthma. J Aerosol Med Pulm Drug Deliv. 2013 Aug;26(4):190-9. doi: 10.1089/jamp.2012.0977. Epub 2012 Oct 25. PMID 23098325